CLINICAL TRIAL: NCT04600713
Title: Physiotherapist Led Exercise Within Cardiac Rehabilitation and Inspiratory Muscle Training and Patients With Paroxysmal Atrial Fibrillation - a Randomized Controlled Trial
Brief Title: Physiotherapist-led Exercise Within Cardiac Rehabilitation and Paroxysmal Atrial Fibrillation and COVID-19.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to logistical problems
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 273293
Record Dates: First submitted 2020-10-09; First posted 2020-10-23 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2023-10

CONDITIONS: Atrial Fibrillation Paroxysmal
Keywords: Health Related Quality of Life; Exercise; Physiotherapy; Physical Activity
MeSH Terms: conditions — Atrial Fibrillation; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized controlled multicenter study
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PT-X and IMT (Experimental): Physiotherapist-led exercise-based cardiac rehabilitation (PT-X) and inspiratory muscle training (IMT).
  Interventions: Other: PT-X and IMT
- Control (No Intervention): The participants in the control group will be offered PT-X at the end of the control period.

INTERVENTIONS:
Other: PT-X and IMT — The intervention consists of PT-X, including central circulatory exercise and muscle exercises, 2 times/week, 60 min/session for 12 weeks, and homebased exercises 2 times/week logged in an exercise diary. For IMT the Threshold Inspiratory Muscle Trainer (Threshold IMT) (Respironics Inc., Murrysville, PA, USA) will be used at 30 % of maximal expiratory pressure in 15 minutes 2 times a day during 12 weeks.
  Arms: PT-X and IMT

SUMMARY:
Paroxysmal atrial fibrillation (AF) induce, in the affected patient, a prominent negative effect on health-related quality of life (HR-QoL) and physical fitness. The health care utilisation is high and the patient does never know when the next attack of atrial fibrillation occurs. Therefore, is physical exertion often avoided due to fear of new attacks. Further, are shortness of breath and fatigue often present despite of prescribed modern drugs. Paroxysmal AF per se enhance markedly the risk to develop stroke and heart failure, which both are syndromes that cause further negative effect on the patient´s HR-QoL and physical fitness. Altogether, cause the symptoms in paroxysmal AF a vicious spiral where both VO2max and muscle function deteriorate. The problems with shortness of breath might be due to dysfunction in respiratory muscles. Physiotherapy led exercise within cardiac rehabilitation (PT-X) in combination with inspiratory muscle training (IMT) has shown positive effects in patients with permanent atrial fibrillation. However, to our knowledge, not yet investigated in patients with paroxysmal AF.

Aim: Primary to investigate, in a multicentre randomised controlled trial, if PT-X in combination with IMT can impact HR-QoL in patients with paroxysmal AF. Secondary to investigate the effect of PT-X in combination with IMT regarding symptoms, physical fitness, physical activity and the number of atrial fibrillation attacks and health care costs compared to the control group, asked to live their usual life, during the study period.

Expected outcome: PTX in combination with IMT can improve HR-QoL, respiratory muscle function, level of symptoms, physical fitness and physical activity in patients with paroxysmal AF. In addition, a reduced number of atrial fibrillation attacks could decrease the direct cost of health care.

DETAILED DESCRIPTION:
Introduction Paroxysmal atrial fibrillation (AF) induce, in the affected patient an increased risk of stroke and heart failure. The corner stone in the medical treatment for AF is anticoagulants and heartrate regulators which affect the physical fitness. Other interventions available for rhythm regulation such as antiarrhythmic drugs, cardioversion and catheter ablation are alternatives aimed to be relief the symptoms of AF and increase the health-related quality of life (HR-QoL). Despite this advanced pharmacologic- and electrotherapy studies evaluating Patient Related Outcomes measures (PROMs) have shown that the symptoms persist and the HR-QoL is still reduced after treatment. Furthermore, Gleason et al, have recently shown that women have a comparatively higher frequency of symptoms, anxiety and depression despite type of intervention. The majority > 90 %, of the patients with paroxysmal AF have symptoms such as palpitations, chest pain, reduced physical fitness and breathlessness. The unpredictability regarding the source of an AF attack, duration and frequencies causes the patient suffering, high healthcare utilization and increased sick leave, this result in high expenditures for AF related causes both for the patient and society. To avoid physical activity and exercise due to fear of an AF attack is not unusual, which may further lead to a reduced physical fitness i.e maximal oxygen capacity (VO2max) and an increased risk of stroke and mortality. This may lead to an evil circle with additional reduced physical fitness, possibly an increase in symptoms and a more reduced HR-QoL. The underlying causes of reduced physical fitness and breathlessness associated with AF is probably multifactorial. One reason could be skeletal muscle abnormities as in heart failure, which often coexists with AF. An increased mortality in the novel Coronavirus (COVID-19) caused by the SARS-CoV-2 is seen in individuals with older age, cardiovascular disease and in men, and the most usual complication is arrythmia such as AF. COVID-19 is a disease that affect the persons lungs and it is not uncommon with pulmonary complications. This can lead to an increased demand for exercise-based rehabilitation in patients with AF and reduced inspiratory muscle strength. One study has shown that a reduced respiratory muscle function can positively be affected with inspiratory muscle training in patients with permanent AF. Furthermore, a Cochrane report have shown that exercise can improve physical fitness in patients with AF, however, no effect was seen in HR-QoL. However, patients with paroxysmal AF, were underrepresented and additional studies concerning patients with paroxysmal AF are requested. Whether physiotherapist-led exercise-based cardiac rehabilitation (PT-X) and inspiratory muscle training (IMT) can improve physical fitness and positively affect symptoms and consequently improve HR-QoL is to our knowledge not studied.

Aim Primary to investigate, in a multicentre randomised controlled trial, if PT-X in combination with IMT can impact HR-QoL in patients with paroxysmal AF. Secondary to investigate the effect of PT-X in combination with IMT regarding symptoms, physical fitness, physical activity and the number of atrial fibrillation attacks and health care costs compared to the control group, asked to live their usual life, during the study period. Further to investigate the prevalence of antibodies for SARS-CoV-2, and the patient's own experience of how COVID-19 has affected their incidence and symptoms of paroxysmal AF.

Question formulations:

Primary question How will participation in PT-X and IMT impact the short form SF-36 general health score compared to the control group that is allowed to continue with their usual life? Secondary questions How will participation in PT-X and IMT impact the exercise capacity compared to the control group that is allowed to continue with their usual life? How will participation in PT-X and IMT affect symptoms of AF and fatigue compared to the control group that is allowed to continue with their usual life? How will participation in PT-X and IMT affect the muscle function compared to the control group that is allowed to continue with their usual life? How will participation in PT-X and IMT affect the frequency, duration and number of AF attacks compared to the control group that is allowed to continue with their usual life? How is the incidence of depression among the participants in the study, and is it possible to impact the prevalence of AF with participation in PT-X and IMT compared to the control group that is allowed to continue with their usual life? How has the COVID-19 affected the patient's own experience of number of attacks, symptoms and duration of AF? How is the prevalence of antibodies for SARs-CoV-2 among the participants in the present study? Method Study design A multi-centre randomised controlled trial Patients A total of 180 patients with paroxysmal AF, age 40 - 85 years, visiting the cardiology clinic at SV Hospital group Alingsås Hospital, Sahlgrenska University Hospital and primary care will be asked to participate in the study. Advertising in the daily press will be made for participants with paroxysmal AF. The patients will be informed both verbal and in written information, and a written informed consent will be obtained.

Statistics and power calculation The patients will be randomised stratified after sex, age and exercise capacity measured by the symptom-limited ergometer cycle test. Ratio and interval data will be presented as mean (± 1 SD), ordinal data will be presented as median (range) and nominal data in absolute and relative numbers. Depending on if the data are normal distributed or not the Student T-Test or the Mann-Whitney U- test will be used for evaluation of differences between the groups. Chi2 test will be used for evaluation of differences between the nominal data.

The sample size was calculated using a power (β) of 80% and a significance level of (α) 5%. Based on the assumption of a mean (SD) significant (p=0.05) difference in the PT-X group compared to the control group regarding improvement of SF-36 General Health score of 7.5 ± 15 points a total of 76 patients are needed in each group. Based on the assumption of a calculated withdraw of approximately 20% a total of 180 participants are needed to be included in this study.

ELIGIBILITY:
Inclusion Criteria:

* Paroxysmal atrial fibrillation verified with electrocardiogram (ECG)
* Left ventricular ejection fraction (EF) ≥ 45% verified by Echocardiography

Exclusion Criteria:

* Ongoing participation in regular aerobic and muscular endurance exercises more than 1 time per week.
* Participation in a weight reduction program.
* Smoking cessation program
* Treatment for sleep apnoea.
* Coronary event or angina pectoris within 3 months prior to inclusion
* stroke with residual symptoms
* presence of pacemaker
* No significant valvular lesions verified by Echocardiography.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The patients are randomized stratified to age, gender and exercise capacity measured by the symptom-limited ergometer cycle test.
Enrollment: 0 (Actual)
Dates: Start 2024-10 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life | Change from baseline at 12 weeks
  The Swedish version of short form 36 (SF-36) will be used for self-reported HR-QoL.

SECONDARY OUTCOMES:
N-terminal pro-B type natriuretic peptide (NT-proBNP) | At baseline
  Venous blood samples will be obtained according to the European accreditation system.
Antibodies for SARS-CoV-2 | At baseline
  Venous blood samples will be obtained investigated with a laboratory method Enzyme- Linked Immunosorbent Assey (ELISA) where antibodies Ig A, Ig G, Ig M will be detected. Due to the fact that the reliability for the laboratory tests to detect antibodies for SARS-CoV-2 is still changing the final decision regarding on which test to use will be made at the start of the study.
Inspiratory and expiratory muscle strength | Change from baseline at 12 weeks
  will be measured with MicroRPM (Micro Medical/Care Fusion, Kent, United Kingdom). The respiratory pressure measures inspiratory and expiratory muscle strength.
Exercise capacity | Change from baseline at 12 weeks
  will be measured by a symptom-limited ergometer cycle test based on World Health Organization (WHO) protocol. The workload begins at 25 W or 50 W depending on the anamnesis. The Watts increase every 4.5 min by 25 W until the patient's rates perceived exertion (RPE) 17 (Very Heavy) on the Borg scale. Unless the patient shows any symptoms or signs that demands an earlier stop at the test. Heart rate and blood pressure are assessed at rest and during the test. If the patient do not surpass the last 4.5 minute the watt will be estimated according to Strandells formula.
Muscle function | Change from baseline at 12 weeks
  will be measured by a muscle endurance test, including the following: A unilateral isoinertial shoulder flexion test assessed with the patient sitting on a stool with their back touching the wall holding a dumbbell in their hand, 2 kg for women and 3 kg for men. The tested arm is elevated to 90º flexion and the arm not tested is placed in the patient's knee. A pace of 40 beats per min is kept by a digital metronome.
  Bilateral isometric shoulder abduction is assessed with the patient holding a 1 kg dumbbell in each hand using the same body position as above. The patient is asked to elevate both arms to 90°of shoulder abduction and to maintain this position as long as possible (measured in s).
  Unilateral isoinertial heel-lift is assessed with the patients performing as many unilateral heel-lifts as possible, with a straight knee, on a 10° tilted wedge, with shoes on. A pace of 60 beats per minutes is kept is kept by a metronome.
Physical activity | Change from baseline at 12 weeks
  will be measured by an accelerometer (Actigraph® GT3x+, Actigraph, Pensacola, Florida, USA). The accelerometer will be worn throughout the whole day during seven days except when taking a bath or a shower. The accelerometer has showed to be valid and reliable in the adult population.
Self reported physical activity | Change from baseline at 12 weeks
  will be measured by short form International Physical Activity Questionnaire (IPAQ). IPAQ measures physical activity during seven days and total time spent sitting a day. IPAQ is validity and reliability tested in several countries.
Self-reported anxiently and depression | Change from baseline at 12 weeks
  will be measured by the Hospital Axiently and Depression Scale (HADS ).
Handheld ECG heart rhythm | Through the study completion, an avarage of 12 weeks
  will be measured with a handheld ECG monitor Zenicor-EKG ® (Zenicor Medical Systems AB, Stockholm, Sverige). Zenicor ® has high specificity and sensitivity for detection of sinus rhythm compared to a 24- Holter ECG. Self- reported AF attacks will be logged in a diary.
Direct hospital costs related to AF | Through the study completion, an avarage of 12 weeks
  are calculated as total costs per patient and the patients medical journal in hospital and primary care.

OTHER OUTCOMES:
Ejection fraction | At baseline
  Will be investigated will be examined during sinus rhythm with a two -dimensional, Doppler echocardiography (Vidid 7 and Vivid E9, GE Medical systems, Horten, Norway).
Left ventricular function | At baseline
  Will be investigated will be examined during sinus rhythm with a two -dimensional, Doppler echocardiography (Vidid 7 and Vivid E9, GE Medical systems, Horten, Norway).
Diastolic function | At baseline
  Will be investigated will be examined during sinus rhythm with a two -dimensional, Doppler echocardiography (Vidid 7 and Vivid E9, GE Medical systems, Horten, Norway).
Valvular screening | At baseline
  Will be investigated will be examined during sinus rhythm with a two -dimensional, Doppler echocardiography (Vidid 7 and Vivid E9, GE Medical systems, Horten, Norway).

CONTACTS AND LOCATIONS:
Overall Officials: Maria Borland, PhD RPT, Principal Investigator — SV Hospital Group, Alingsås hospital Sweden

REFERENCES:
- [Background] Kirchhof P, Benussi S, Kotecha D, Ahlsson A, Atar D, Casadei B, Castella M, Diener HC, Heidbuchel H, Hendriks J, Hindricks G, Manolis AS, Oldgren J, Popescu BA, Schotten U, Van Putte B, Vardas P, Agewall S, Camm J, Baron Esquivias G, Budts W, Carerj S, Casselman F, Coca A, De Caterina R, Deftereos S, Dobrev D, Ferro JM, Filippatos G, Fitzsimons D, Gorenek B, Guenoun M, Hohnloser SH, Kolh P, Lip GY, Manolis A, McMurray J, Ponikowski P, Rosenhek R, Ruschitzka F, Savelieva I, Sharma S, Suwalski P, Tamargo JL, Taylor CJ, Van Gelder IC, Voors AA, Windecker S, Zamorano JL, Zeppenfeld K. 2016 ESC Guidelines for the management of atrial fibrillation developed in collaboration with EACTS. Europace. 2016 Nov;18(11):1609-1678. doi: 10.1093/europace/euw295. Epub 2016 Aug 27. No abstract available. PMID 27567465
- [Background] Hobbs FD, Kenkre JE, Roalfe AK, Davis RC, Hare R, Davies MK. Impact of heart failure and left ventricular systolic dysfunction on quality of life: a cross-sectional study comparing common chronic cardiac and medical disorders and a representative adult population. Eur Heart J. 2002 Dec;23(23):1867-76. doi: 10.1053/euhj.2002.3255. PMID 12445536
- [Background] Zhang L, Gallagher R, Neubeck L. Health-related quality of life in atrial fibrillation patients over 65 years: A review. Eur J Prev Cardiol. 2015 Aug;22(8):987-1002. doi: 10.1177/2047487314538855. Epub 2014 Jun 12. PMID 24924742
- [Background] Gleason KT, Dennison Himmelfarb CR, Ford DE, Lehmann H, Samuel L, Jain S, Naccarelli G, Aggarwal V, Nazarian S. Association of sex and atrial fibrillation therapies with patient-reported outcomes. Heart. 2019 Nov;105(21):1642-1648. doi: 10.1136/heartjnl-2019-314881. Epub 2019 May 22. PMID 31118198
- [Background] Dorian P, Jung W, Newman D, Paquette M, Wood K, Ayers GM, Camm J, Akhtar M, Luderitz B. The impairment of health-related quality of life in patients with intermittent atrial fibrillation: implications for the assessment of investigational therapy. J Am Coll Cardiol. 2000 Oct;36(4):1303-9. doi: 10.1016/s0735-1097(00)00886-x. PMID 11028487
- [Background] Hansson A, Madsen-Hardig B, Olsson SB. Arrhythmia-provoking factors and symptoms at the onset of paroxysmal atrial fibrillation: a study based on interviews with 100 patients seeking hospital assistance. BMC Cardiovasc Disord. 2004 Aug 3;4:13. doi: 10.1186/1471-2261-4-13. PMID 15291967
- [Background] Ericson L, Bergfeldt L, Bjorholt I. Atrial fibrillation: the cost of illness in Sweden. Eur J Health Econ. 2011 Oct;12(5):479-87. doi: 10.1007/s10198-010-0261-3. Epub 2010 Jul 1. PMID 20593297
- [Background] Rohrbacker NJ, Kleinman NL, White SA, March JL, Reynolds MR. The burden of atrial fibrillation and other cardiac arrhythmias in an employed population: associated costs, absences, and objective productivity loss. J Occup Environ Med. 2010 Apr;52(4):383-91. doi: 10.1097/JOM.0b013e3181d967bc. PMID 20357675
- [Background] Rienstra M, Lubitz SA, Mahida S, Magnani JW, Fontes JD, Sinner MF, Van Gelder IC, Ellinor PT, Benjamin EJ. Symptoms and functional status of patients with atrial fibrillation: state of the art and future research opportunities. Circulation. 2012 Jun 12;125(23):2933-43. doi: 10.1161/CIRCULATIONAHA.111.069450. No abstract available. PMID 22689930
- [Background] Hussain N, Gersh BJ, Gonzalez Carta K, Sydo N, Lopez-Jimenez F, Kopecky SL, Thomas RJ, Asirvatham SJ, Allison TG. Impact of Cardiorespiratory Fitness on Frequency of Atrial Fibrillation, Stroke, and All-Cause Mortality. Am J Cardiol. 2018 Jan 1;121(1):41-49. doi: 10.1016/j.amjcard.2017.09.021. Epub 2017 Nov 13. PMID 29221502
- [Background] Ueshima K, Myers J, Ribisl PM, Morris CK, Kawaguchi T, Liu J, Froelicher VF. Exercise capacity and prognosis in patients with chronic atrial fibrillation. Cardiology. 1995;86(2):108-13. doi: 10.1159/000176850. PMID 7728799
- [Background] Okita K, Kinugawa S, Tsutsui H. Exercise intolerance in chronic heart failure--skeletal muscle dysfunction and potential therapies. Circ J. 2013;77(2):293-300. doi: 10.1253/circj.cj-12-1235. Epub 2013 Jan 19. PMID 23337207
- [Background] Santhanakrishnan R, Wang N, Larson MG, Magnani JW, McManus DD, Lubitz SA, Ellinor PT, Cheng S, Vasan RS, Lee DS, Wang TJ, Levy D, Benjamin EJ, Ho JE. Atrial Fibrillation Begets Heart Failure and Vice Versa: Temporal Associations and Differences in Preserved Versus Reduced Ejection Fraction. Circulation. 2016 Feb 2;133(5):484-92. doi: 10.1161/CIRCULATIONAHA.115.018614. Epub 2016 Jan 8. PMID 26746177
- [Background] Guzik TJ, Mohiddin SA, Dimarco A, Patel V, Savvatis K, Marelli-Berg FM, Madhur MS, Tomaszewski M, Maffia P, D'Acquisto F, Nicklin SA, Marian AJ, Nosalski R, Murray EC, Guzik B, Berry C, Touyz RM, Kreutz R, Wang DW, Bhella D, Sagliocco O, Crea F, Thomson EC, McInnes IB. COVID-19 and the cardiovascular system: implications for risk assessment, diagnosis, and treatment options. Cardiovasc Res. 2020 Aug 1;116(10):1666-1687. doi: 10.1093/cvr/cvaa106. PMID 32352535
- [Background] Ariansen I, Edvardsen E, Borchsenius F, Abdelnoor M, Tveit A, Gjesdal K. Lung function and dyspnea in patients with permanent atrial fibrillation. Eur J Intern Med. 2011 Oct;22(5):466-70. doi: 10.1016/j.ejim.2011.06.010. Epub 2011 Jul 12. PMID 21925054
- [Background] Risom SS, Zwisler AD, Johansen PP, Sibilitz KL, Lindschou J, Gluud C, Taylor RS, Svendsen JH, Berg SK. Exercise-based cardiac rehabilitation for adults with atrial fibrillation. Cochrane Database Syst Rev. 2017 Feb 9;2(2):CD011197. doi: 10.1002/14651858.CD011197.pub2. PMID 28181684
- [Background] Sullivan M, Karlsson J, Ware JE Jr. The Swedish SF-36 Health Survey--I. Evaluation of data quality, scaling assumptions, reliability and construct validity across general populations in Sweden. Soc Sci Med. 1995 Nov;41(10):1349-58. doi: 10.1016/0277-9536(95)00125-q. PMID 8560302
- [Background] Exercise tests in relation to cardiovascular function. Report of a WHO meeting. World Health Organ Tech Rep Ser. 1968;388:1-30. No abstract available. PMID 4968942
- [Background] STRANDELL T. CIRCULATORY STUDIES ON HEALTHY OLD MEN. WITH SPECIAL REFERENCE TO THE LIMITATION OF THE MAXIMAL PHYSICAL WORKING CAPACITY. Acta Med Scand Suppl. 1964;414:SUPPL 414:1-44. No abstract available. PMID 14161322
- [Background] Borg G. Borg's perceived exertion and pain scales. Leeds: Human Kinetics; 1998.
- [Background] Cider A, Carlsson S, Arvidsson C, Andersson B, Sunnerhagen KS. Reliability of clinical muscular endurance tests in patients with chronic heart failure. Eur J Cardiovasc Nurs. 2006 Jun;5(2):122-6. doi: 10.1016/j.ejcnurse.2005.10.001. Epub 2005 Oct 28. PMID 16257580
- [Background] Doliwa PS, Frykman V, Rosenqvist M. Short-term ECG for out of hospital detection of silent atrial fibrillation episodes. Scand Cardiovasc J. 2009 Jun;43(3):163-8. doi: 10.1080/14017430802593435. PMID 19096977
- [Background] Hendrikx T, Rosenqvist M, Wester P, Sandstrom H, Hornsten R. Intermittent short ECG recording is more effective than 24-hour Holter ECG in detection of arrhythmias. BMC Cardiovasc Disord. 2014 Apr 1;14:41. doi: 10.1186/1471-2261-14-41. PMID 24690488
- [Background] Aadland E, Ylvisaker E. Reliability of the Actigraph GT3X+ Accelerometer in Adults under Free-Living Conditions. PLoS One. 2015 Aug 14;10(8):e0134606. doi: 10.1371/journal.pone.0134606. eCollection 2015. PMID 26274586
- [Background] Van Remoortel H, Giavedoni S, Raste Y, Burtin C, Louvaris Z, Gimeno-Santos E, Langer D, Glendenning A, Hopkinson NS, Vogiatzis I, Peterson BT, Wilson F, Mann B, Rabinovich R, Puhan MA, Troosters T; PROactive consortium. Validity of activity monitors in health and chronic disease: a systematic review. Int J Behav Nutr Phys Act. 2012 Jul 9;9:84. doi: 10.1186/1479-5868-9-84. PMID 22776399
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Polikandrioti M, Koutelekos I, Vasilopoulos G, Gerogianni G, Gourni M, Zyga S, Panoutsopoulos G. Anxiety and Depression in Patients with Permanent Atrial Fibrillation: Prevalence and Associated Factors. Cardiol Res Pract. 2018 Feb 19;2018:7408129. doi: 10.1155/2018/7408129. eCollection 2018. PMID 29670767
- See also: World Health Organization. WHO guidelines on drawing blood — http://apps.who.int/iris/bitstream/10665/44294/1/9789241599221_eng.pdf